CLINICAL TRIAL: NCT06768112
Title: Adaptive Changes in Plasticity of Cerebrum and Cerebellum Following Innovative Postural
Brief Title: Non-Invasive Vagus Nerve Stimulation Combine Postural Training in the Elderly
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NSTC 113-2314-B-006 -080 -MY3
Record Dates: First submitted 2024-09-12; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-09

CONDITIONS: Balanced; Aging
Keywords: Gual-task; Invasive cervical vagus nerve stimulation; Aging; Cerebellar EEG
MeSH Terms: interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): participants in this arm will conduct balance training without non-invasive vagal nerve stimulation.
  Interventions: Behavioral: balance training; Behavioral: Mini-Mental State Examination
- non-invasive vagal nerve stimulation (Experimental): Participants will receive non-invasive vagal nerve stimulation and balance training
  Interventions: Device: Non-Invasive Vagus Nerve Stimulation; Behavioral: balance training; Behavioral: Mini-Mental State Examination

INTERVENTIONS:
Device: Non-Invasive Vagus Nerve Stimulation — Using non-invasive vagus nerve stimulation at the ear to stimulate the adrenergic and serum hormone pathways, activating the frontal lobe system, sensory-motor nervous system, and cerebellum, to investigate the effects and neural mechanisms of dynamic posture training and learning.
  Arms: non-invasive vagal nerve stimulation
Behavioral: balance training — Participants will be asked to stand on a soft-platform and hit on blaze-pod LED within 60 seconds.
Behavioral: Mini-Mental State Examination — The mini-mental state examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment.

SUMMARY:
This three-year research proposal aims to enhance postural control in older adults using non-invasive vagus nerve stimulation (nVNS). The study will develop a new system integrating cerebellar EEG (ECeG), EEG, and ECG to assess how nVNS combined with postural training affects individuals with early-stage frontal degeneration.

In the first year, the focus will be on creating and validating the ECeG system to explore neural mechanisms of postural control. The second year will test the combined effects of ear-nVNS and dynamic posture training, examining how nVNS influences adrenal and hormone pathways. The final year will evaluate if ear-nVNS can further improve postural training with virtual feedback.

Overall, the project aims to advance fall prevention strategies for older adults by exploring the role of cerebellar function and innovative training methods.

DETAILED DESCRIPTION:
The interaction between the cortex and cerebellum is pivotal in adapting to diverse postural challenges. Non-invasive vagus nerve stimulation (nVNS) has recently gained attention as a therapeutic approach with potential effects on frontal facilitation and improvement of neuromotor control. It provides a promising avenue to aid postural training for older individuals experiencing early-stage frontal degeneration. This three-year proposal aims to develop an integrated electrophysiological system for cerebellar EEG (ECeG), EEG, and ECG measures, with the goal of investigating the effects of innovative postural training with nVNS on older adults, particularly those at risk of falls due to frontal aging. The primary focus will be on the reorganization of cortical networks, the functional coupling between the cortex and cerebellum, and heart rate variability, with a contextual extension to the neurovisceral integrative model. In the first year, the proposal seeks to develop and validate a cerebellar electroencephalogram (ECeG) system, integrating it with the EEG and electrocardiogram (ECG) systems to explore the neural mechanisms for postural control on varying stance configurations for the elderly. During the second year, the proposal will investigate the effectiveness and neural mechanisms of combined ear-nVNS and dynamic posture training for the elderly, utilizing the Mesocircuit model to trigger adrenal and serum hormone pathways with nVNS. In the third year, the proposal will examine whether ear-nVNS can further enhance the postural training effects of virtual error amplification feedback in dynamic posture training for the elderly. The highlights of this project include the novel application of ear-nVNS to counteract falls in the elderly due to frontal degeneration and cognitive decline, as well as pioneering approaches to explore neural mechanisms underlying postural training effects with an in vivo examination of the cerebellar role. The innovative postural training with convenience is expected to be of practical value for fall prevention in the elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Participants aged 18-45 years (young adults) and 60-80 years (older adults).
2. Vision should be within the normal range after visual correction.
3. Lower limb strength requirement: Ability to climb stairs without holding onto anything, able to ascend 15 steps (a typical office building floor has approximately 15-20 steps).
4. No history of falls in the past six months.

Exclusion Criteria:

Here is the translation of the provided text:

1. Young adult participants: Exclude students from the Department of Physical Therapy, School of Medicine, and Institute of Behavioral Medicine at National Cheng Kung University.
2. Uncontrolled cardiovascular diseases (e.g., hypertensive patients with resting systolic blood pressure exceeding 160 mmHg).
3. Lower limb venous embolism, arterial calcification, and lymphatic issues.
4. Diabetes, sickle cell anemia, coagulation disorders, dialysis patients, and those with conditions affecting walking, lower limb musculoskeletal function, and balance issues.
5. No known psychiatric, neuromuscular, or degenerative neurological diseases.
6. Hearing impairment or those using hearing aids.
7. Dizziness caused by any lesions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive Performance | the first day, at the end of 5 days training
  Analysis of cognitive tests including Stroop test and trail making test.
Brain activity | the first day, at the end of 5 days training
  EEG Data Analysis
Kinematic Analysis of Upper and Lower Limb Dynamics | the first day, at the end of 5 days training
  Participants are asked to stand with both feet on a soft-pad and try to maintain a stable posture with minimal body sway. The center of pressure trajectory are taken to estimate behavioral and neurophysiological mechanisms. The dual-task involves performing simultaneous tasks of tapping LED sensor lights in real-time while standing on the soft-pad force plate.

OTHER OUTCOMES:
Mini-Mental State Examination; MMSE | Before participating in the formal protocol, each subject must take the Mini-Mental State Examination to assess their cognitive level. This test is conducted only once per subject.
  A total score of 30 points; a score below 24 indicates mild cognitive impairment. Those with mild impairment will be evenly distributed into groups.

CONTACTS AND LOCATIONS:
Locations (1):
- National Chen Kong University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No